CLINICAL TRIAL: NCT07168746
Title: National Cohort of Patients With SITRAME Syndrome
Acronym: CO-SITRAME
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250008
Record Dates: First submitted 2025-06-17; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Auto Inflammatory Diseases
Keywords: SITRAME; autoinflammatory diseases; cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SITRAME syndrome is a recently described disease. In the absence of epidemiological data on SITRAME syndrome in France, the National Reference Center for Autoinflammatory Diseases proposes coordinating a database to collect both retrospective and prospective cases of this rare disease.

Currently, there are no available data on the epidemiology or treatment of SITRAME syndrome in France or globally. The importance of this research is to provide an overview of demographic, etiological, and disease progression data for patients with SITRAME syndrome in France. This will allow the establishment of quantitative data on the morbidity and mortality of this rare disease.

ELIGIBILITY:
Inclusion Criteria:

• SITRAME syndrome meeting the diagnostic criteria for the disease

All the following criteria must be met:

1. Systemic inflammation: at least 1 documented episode of CRP >5mg/mL during a skin flare
2. Maculopapular rash on the trunk: fixed, non-itchy maculopapular rash on the trunk appearing within hours with clear borders
3. Recurrence in the same areas: at least 3 different episodes
4. Acute: duration less than 8 days

And at least 1 of the following criteria:

1. Fever during flare-ups
2. Flare-ups triggered by infections, vaccinations, or intense physical exercise
3. Fatigue during and/or after flare-ups
4. Associated papular rash

And all the following exclusion criteria must be met:

* No evidence of a monogenic autoinflammatory disease, evolving neoplasm, or evolving autoimmune disease.
* Adult patients at the time of inclusion
* Patients not opposed to participating in the research

Exclusion Criteria:

- Persons with special protection cannot be included in the study:

* Adults under guardianship or curatorship
* Hospitalized persons without consent and not legally protected
* Persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in France via the national reference center for autoinflammatory diseases at Tenon Hospital (Internal Medicine, Dermatology and Allergology Department at Tenon Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2055-09 (Estimated)

PRIMARY OUTCOMES:
Description of the sexe at the diagnosis of the disease in order to describe the clinical characteristics of patients followed for SITRAME syndrome | Day 0- Baseline
Description of the age at the diagnosis of the disease | Day 0- Baseline
  Description of the age at the diagnosis of the disease in order to describe the clinical characteristics of patients followed for SITRAME syndrome
Description of cardiovascular co-morbidity | Day 0- Baseline
  Description of cardiovascular co-morbidity at the diagnosis of the disease in order to describe the clinical characteristics of patients followed for SITRAME syndrome
Description of presence of an allergical context | Day 0- Baseline
  Description of presence of an allergical context in order to describe the clinical characteristics of patients followed for SITRAME syndrome
Description of the different therapeutic lines | Year 15
  Description of the different therapeutic lines in order to describe the clinical characteristics of patients followed for SITRAME syndrome
Description of the age at death | Day 0- Baseline
  Description of the age at death in order to describe the clinical characteristics of patients followed for SITRAME syndrome

SECONDARY OUTCOMES:
Measure of the prevalence of this disease annually using the register of newly included patients | Every year up to 15 years
Measure of the incidence of this disease | Every year up to 15 years
  Measure of the incidence of this disease annually using the register of newly included patients Time frame: annually
Description of the rare clinical manifestations (outside of the well-established disease criteria) | Year 15
Description of the rare biological manifestations (outside of the well-established disease criteria) | Year 15
Measure of the number of patients eligible for various clinical research studies on SITRAME syndrome | Every year up to 15 years
Measure of the proportion of patients using targeted therapies throughout the study | Year 15
Measure of the number of deaths in patients followed for SITRAME syndrome | every 5 years up to 15 years
Description of the death causes in patients followed for SITRAME syndrome | every 5 years up to 15 years
Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (pulmonary manifestations) | every 5 years up to 15 years
  Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (pulmonary manifestations) in order to describe the clinical characteristics of this population
Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (cardiac manifestations) | Every 5 years up to 15 years
  Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (cardiac manifestations) in order to describe the clinical characteristics of this population
Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (neurological manifestations) | every 5 years up to 15 years
  Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (neurological manifestations) in order to describe the clinical characteristics of this population
Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (gastrointestinal manifestations) | every 5 years up to 15 years
  Number of dead patients followed for SITRAME syndrome with presence and pattern of extracutaneous involvement (gastrointestinal manifestations) in order to describe the clinical characteristics of this population
C-reactive protein (CRP) rate in the population of dead patients followed for SITRAME syndrome | every 5 years up to 15 years
  C-reactive protein (CRP) rate in the population of dead patients followed for SITRAME syndrome in order to describe the biological characteristics of this population
Frequency of inflammatory flares throughout the disease course in the population of dead patients followed for SITRAME syndrome | every 5 years up to 15 years
  Frequency of inflammatory flares throughout the disease course in the population of dead patients followed for SITRAME syndrome in order to describe the biological characteristics of this population
Ferritin rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Ferritin rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Liver enzymes rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Liver enzymes rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Creatinine rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Creatinine rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Red blood cells rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Red blood cells rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Platelets rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Platelets rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Hemoglobin rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Hemoglobin rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Hematocrit rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Hematocrit rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Mean corpuscular volume (MCV) rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Mean corpuscular volume (MCV) rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
White blood cells rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  White blood cells rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Neutrophils rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Neutrophils rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Lymphocytes rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Lymphocytes rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Monocytes rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Monocytes rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Eosinophils rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Eosinophils rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population
Basophils rate of the dead patient followed for SITRAME syndrome | every 5 years up to 15 years
  Basophils rate of the dead patient followed for SITRAME syndrome in order to describe the biological characteristics of this population

CONTACTS AND LOCATIONS:
Overall Officials: Angele SORIA, PUPH, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No